CLINICAL TRIAL: NCT03285165
Title: Cerebral Vascular Effects of Dexmedetomidine Versus Propofol Sedation in Intubated Mechanically Ventilated ICU Patients With and Without Traumatic Brain Injury.
Brief Title: Cerebral Vascular Effects of Dexmedetomidine Versus Propofol Sedation in Intubated Mechanically Ventilated ICU Patients
Acronym: DEXSEDATION
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: NO AVAILABLE FUND
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200002
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: this study will be accomplished to investigate the effect of dexmedetomidine sedation on the cerebral blood flow in intubated mechanically ventilated trauma patients with and without traumatic brain injury, in comparison with propofol.
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DEX I (Active Comparator): Trauma Patients without TBI received 0.2-0.7 mcg/kg/h dexmedetomedine infusion.
  Interventions: Drug: 0.2-0.7 mcg/kg/h dexmedetomedine infusion.
- DEX II (Active Comparator): Trauma Patients with TBI received 0.2-0.7 mcg/kg/h dexmedetomedine infusion.
  Interventions: Drug: 0.2-0.7 mcg/kg/h dexmedetomedine infusion.
- Propofol I (Active Comparator): Trauma Patients without TBI received 10-70 mcg/kg/h propofol infusion.
  Interventions: Drug: 10-70 mcg/kg/h propofol infusion.
- Propofol II (Active Comparator): Trauma Patients with TBI received 10-70 mcg/kg/h propofol infusion.
  Interventions: Drug: 10-70 mcg/kg/h propofol infusion.

INTERVENTIONS:
Drug: 0.2-0.7 mcg/kg/h dexmedetomedine infusion. — patients will receive dexmedetomidine 0.2-0.7 mcg/kg/h infusion for 24h.
  Other Names: Precedex
  Arms: DEX I; DEX II
Drug: 10-70 mcg/kg/h propofol infusion. — Patients will receive 10-70 mcg/kg/h propofol infusion for 24h.
  Other Names: Deprivan
  Arms: Propofol I; Propofol II

SUMMARY:
Serial transcranial Doppler (TCD) exams in healthy volunteers and in animal models showed a strong linear relationship between middle cerebral artery (MCA) flow velocity (FV) and dexmedetomidine infusion. The concomitant elevation of pulsatility index (PI) indicates vasoconstriction of the cerebral vasculature as the most profound underlying mechanism.

DETAILED DESCRIPTION:
Available clinical evidence on the use of dexmedetomidine sedation in neurosurgical and neurocritical care is limited and no definite conclusion can be drawn. There is a need for The use of dexmedetomidine might be a useful adjunct in clinical situations when the increase in CBF could be detrimental such as vasogenic cerebral edema (i.e., TBI, large brain tumors). However, dexmedetomidine sedation is questionable in patients with subarachnoid hemorrhage and acute stroke, since the associate drop in arterial pressure could worsen the coexisting increase in circulating catecholamines and massive sympathetic outflow. Further high-quality RCTs to evaluate the use of dexmedetomidine as a sedative agent both in general ICU patients and in patients with TBI.

Transcranial Doppler (TCD) is a simple noninvasive bedside tool to assess the cerebral blood flow pattern. The new development of transcranial color Doppler with angle correction option helps to improve the sensitivity of test results. TCD can assess the evolution of CBF alterations and possibly cerebral autoregulation performance and ICP estimation in patients presenting with cerebral pathology.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients (18-50 years old, ASA I-II).
* With and without mild TBI.
* Mild traumatic brain injury will include; brain edema, brain contusion, fracture base, fissure fracture and depressed fracture.
* The severity of traumatic brain injury will be defined as mild based on basal Glasgow Coma Scale and basal Computerized tomography scanning.
* Requirements of endotracheal intubation, mechanical ventilation and light to moderate sedation because of associated abdominal or chest traumatic injuries.
* The sedation needed should of an estimated duration not less than 24h.
* Baseline hemodynamic parameters within the normal range.
* Baseline middle cerebral artery flow velocity within the normal range.

Exclusion Criteria:

* Severe traumatic brain injury, subarachnoid hemorrhage and Intra-cerebral hemorrhage.
* Spinal cord injury.
* Hemodynamically unstable patients and patients on inotropes.
* Patients who have a cardiac pacemaker or automatic implantable cardioverter defibrillator.
* Patients with hepatic or renal impairment.
* Pregnant females.
* Patients who are incarcerated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2021-09-16 (Estimated); Study Completion 2021-09-16 (Estimated)

PRIMARY OUTCOMES:
Middle cerebral artery flow velocity | 24 hours
  1. Right and left middle cerebral artery (MCA) will be measured via trans-temporal window and the depth of insinuation will be between 30-60 mm with the subject's head in neutral position. Mean values of simultaneously measured invasive blood pressure recordings and the outer envelope of time averaged MCA flow velocity (FV) recordings during ten consecutive cardiac cycles

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- Assiut university main hospital, Trauma ICU, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No